CLINICAL TRIAL: NCT01908569
Title: Application of MACS (Magnetic-activated Cell Sorting) and Time-lapse Technology (Embryoscope) in Assisted Reproduction Patients With Good Prognosis
Brief Title: Application of MACS and Time-lapse Technology in Good-prognosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IVISEV-004ROVIC
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: MACS Technique Efficacy
Keywords: MACS, time-lapse, embryo, spermatozoid, sperm

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- NO MACS + Time-lapse technology (Active Comparator): The sperm capacitation will be performed through a density gradient. This sperm will be used in the IVF/ICSI treatment of the patient and the embryos obtained will be cultured using time-lapse technology (Embryoscope).
  Interventions: Other: NO MACS
- MACS + time-lapse technology (Experimental): The sperm capacitation will be performed through a density gradient. After that, it will be subjected to the MACS technique in order to select the non-apoptotic spermatozoids. This sperm will be used in the IVF/ICSI treatment of the patient and the embryos obtained will be cultured using time-lapse technology (Embryoscope).
  Interventions: Other: MACS

INTERVENTIONS:
Other: MACS — The sperm will be subjected to capacitation through a density gradient together with the MACS technique in order to select the non-apoptotic spermatozoids.
  Arms: MACS + time-lapse technology
Other: NO MACS — The sperm capacitation will be performed through a density gradient. The MACS technique will not be applied.
  Arms: NO MACS + Time-lapse technology

SUMMARY:
The MACS technique (magnetic-activated cell sorting) is based on the usage of microbeads, magnetic particles with a diameter of 35 nanometers joined to the compound annexin V. Annexin V is a protein with a high affinity for the molecule phosphatidylserine. This system allow us to eliminate those spermatozoids which have begun the apoptosis and have phosphatidylserine residues on their membrane surface. Using this technique, the apoptotic spermatozoids will join the microbeads and consequently be retained in a column applying a magnetic field.

Recent studies show the benefits of spermatozoid selection using MACS and the improvement in mobility, viability, DNA fragmentation and fertilization potential. It has also been observed an improvement in the embryo cells division rate, clinical pregnancy rates and spermatozoid survival after thawing. However, it is necessary to perform new clinical studies in order to evaluate the real potential of this technology and its safety.

The purpose of this study is to evaluate the effect of the MACS technique on the clinical results of good-prognosis patients who are going through IVF/ICSI treatments in order to achieve a pregnancy.

The hypothesis of this study is that the application of the MACS technique in assisted reproduction treatments is associated with a better embryo quality and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* <38 years
* >10 follicles with a diameter of ≥10 mm the day before the follicular puncture

Exclusion Criteria:

* Patients subject to preimplantation genetic diagnosis treatments

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 14 months

SECONDARY OUTCOMES:
Pregnancy rate | 14 months
Embryo quality | 14 months
  According to ASEBIR criteria
Implantation rate | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor Blasco, MSc, Study Chair — Vida Recoletas Sevilla; Rocío Quiroga, MSc, Principal Investigator — Vida Recoletas Sevilla; Cristina González, PhD, Study Chair — Vida Recoletas Sevilla; Cinzia Caligara, MD, Study Chair — Vida Recoletas Sevilla
Locations (1):
- IVI Sevilla, Seville, Spain